CLINICAL TRIAL: NCT02996240
Title: A Phase 0, Investigator Initiated Study, Evaluating the Impact of Omega 3 Free Fatty Acid Supplementation on Breast Cancer (CTMS# 16-0119)
Brief Title: Breast, Omega 3 Free Fatty Acid, Ph 0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Virginia G. Kaklamani, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 16-0119; 16-665H (Other: UTHSCSA)
Record Dates: First submitted 2016-12-12; First posted 2016-12-19 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Breastcancer
MeSH Terms: interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Omega-3 FFA (Experimental): Patients will take 12 capsules daily with meals, divided twice daily (example, 6 with breakfast and 6 with dinner).
  Interventions: Dietary Supplement: Omega-3 FFA

INTERVENTIONS:
Dietary Supplement: Omega-3 FFA — Omega-3 Free Fatty Acid will be given as a fish oil in a capsule.
  Other Names: Omacor

SUMMARY:
Assess the impact of dietary omega 3 free fatty acids breast cancer patients.

DETAILED DESCRIPTION:
Prospective, single arm, short term study with correlative biomarker endpoints. Two hundred (200) newly diagnosed breast cancer patients will be recruited to participate in a short term (30 day) Phase 0 biomarker evaluation study prior to surgical resection. Patients will be receive fish Oil (Omega-3 FFAs, 2700 mg by mouth twice daily).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* ECOG ≤2
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Consented for tissue collection on CTRC repository 07-32

Exclusion Criteria:

* Active systemic illness (infection including viral illnesses such as Hepatitis and HIV)
* Chronic use of NSAIDs or omega-3 free fatty acid supplementation within the last 60 days (defined as greater than or equal to 7 consecutive days)
* Any NSAIDs or omega-3 free fatty acid supplementation within the last 14 days
* History of medical noncompliance
* Scheduled date of surgical resection that would limit the amount of time taking the intervention to less than 21 days

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Change in serum colony stimulating factor at surgery | 30 days
Change in circulating levels of pro-inflammatory cytokines. | 30 days
Change in circulating levels of eicosanoids. | 30 days
Change in circulating levels of metabolics. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Virginia G Kaklamani, MD, Principal Investigator — Principal Investigator
Locations (1):
- CTRC at University of Texas Health Science Center San Antonio, San Antonio, Texas, United States